CLINICAL TRIAL: NCT02008409
Title: Evaluation of Safety and Efficacy of the EndoLift Liver Retractor: a Pilot Study of a New Internal Laparoscopic Liver Retraction Device
Brief Title: Evaluation of Safety and Efficacy of the EndoLift Liver Retractor
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated. Six subjects were consented & all were withdrawn before any study activities took place.
Sponsor: Duke University (Other)
Collaborators: Virtual Ports (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00028255
Record Dates: First submitted 2013-11-22; First posted 2013-12-11 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: Minimally Invasive Surgical Procedure; Laparoscopic Gastric Banding; Laparoscopic Roux-en-Y Gastric Bypass; Laparoscopic Sleeve Gastrectomy; Laparoscopic Fundoplication Procedure; Laparoscopic Heller Myotomy; Laparoscopic Paraesophageal Hernia Repair; Laparoscopic Gastric Resection
Keywords: Minimally Invasive Surgery; EndoLift Liver Retractor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EndoLift Liver Retractor (Experimental): During surgery, the surgeon will use the new internal liver retractor device. The device will retract the subject's liver out of the way and help the surgeon see better during the surgery. The device is placed inside the abdomen during the surgery. It is "clipped" onto 2 safe surfaces inside the abdomen. The device is removed before the surgery ends.
  Interventions: Device: EndoLift Liver Retractor

INTERVENTIONS:
Device: EndoLift Liver Retractor — During the surgery, the surgeon will use the new internal liver retractor device. The device will retract the liver out of the way and help the surgeon see better during the surgery. The device is placed inside the abdomen during the surgery. It is "clipped" onto 2 safe surfaces inside the abdomen. The device is removed before the surgery ends.

SUMMARY:
The primary goal of the study is to evaluate the safety of the EndoLift Liver Retractor as an internal laparoscopic liver retraction device. The secondary goals of the study are to evaluate the efficacy of the EndoLift Liver Retractor as an internal laparoscopic liver retraction device and to identify 'best practices' for device utilization.

This study evaluates the use of a specific type of liver retractor (EndoLift). Liver retractors are often necessary during MIS procedures, but this retractor is the only device which is deployed internally (NOT requiring additional skin punctures/incisions for placement of the liver retractor device). All patients undergoing minimally invasive surgery (MIS) at Duke Regional Hospital will be approached.

The new device is expected to have a minimal risk safety profile. The investigators believe that these risks are no more than would be encountered by using any other commercially available retraction device available on the market today. Data will be collected and analyzed by the identified investigators. Continuous variables will be analyzed via T-test and Chi-square analysis will be applied to discontinuous variables. Statistical analysis software such as SPSS® will be utilized when necessary.

DETAILED DESCRIPTION:
Since the introduction of minimally invasive surgery (MIS) techniques in the 1980's laparoscopic surgery has become the preferred approach for a number of intra-abdominal procedures such as cholecystectomy, gastric bypass, etc.[1] One of the key components of laparoscopic surgery, of any surgery for that matter, is the ability to achieve and maintain adequate visualization of the surgical target throughout the procedure. During certain MIS procedures the patient's internal organs, such as the liver, can block or obscure the surgical view. A number of surgical instruments (retractors) have been developed to help retract abdominal organs "out of the way" during MIS procedures, but all of these devices require an additional abdominal wall puncture/incision to adequately position the device.

Virtual Ports, Ltd. has developed a new laparoscopic liver retractor device, the EndoLift Liver Retractor. This new device does not require additional skin incisions and is placed internally (inside the abdomen) during laparoscopic surgery. The device has 2 ends that "grab" tissue. The body of the device is a smooth, cylindrical steel bar that has minimal risk of traumatizing tissues/organs. The ends of the device are positioned on to peritoneal surfaces (e.g., anterior abdominal wall and/or the right crus of the diaphragm) and the body of the device (smooth cylindrical bar) "pushes" the liver away from the surgical field.

ELIGIBILITY:
Inclusion Criteria:

Subjects eligible for this clinical study must fulfill all of the following:

* Subject is 18 years of age or older.
* Subject is scheduled for a MIS procedure:

  1. Laparoscopic Gastric Banding
  2. Laparoscopic Roux-en-Y Gastric Bypass
  3. Laparoscopic Sleeve Gastrectomy
  4. Laparoscopic Fundoplication Procedure (Nissen, Toupet, Dor, etc.)
  5. Laparoscopic Heller myotomy
  6. Laparoscopic paraesophageal hernia repair
  7. Laparoscopic gastric resection
* Subject is able to comprehend and give informed consent for participation in this study.

Exclusion Criteria:

* Subjects not eligible for this research study include those that have any of the following:

  * Subject is unable to comprehend and give informed consent for participation in this study.
  * Subject who are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-11; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Safety | Day 1 post-op
  The primary study endpoint will be to establish the safety of using the EndoLift Liver Retractor as an internal laparoscopic liver retraction device.
  Safety will be established by lack of serious events. Events are defined as adverse if they require change in the operative course, a device specific complication and/or association with prolongation of hospital stay.

SECONDARY OUTCOMES:
Effective use of the EndoLift Liver Retractor | Up to 6 hours during the operative procedure
  The effective use of the EndoLift Liver Retractor as a liver retraction device during surgery will be considered a "success". If there is a need to use any additional equipment to retract the liver during the surgery, the subject will be scored a "failure".
  Study success will be declared if at least 80% of subjects are scored a "success".

OTHER OUTCOMES:
Physician satisfaction | Day 1 Post-op
  Physician satisfaction and surgeon recommendations for 'best practices' during utilization of the EndoLift Liver Retractor will be assessed by questionnaire.
  Study outcomes will be measured within the hospitalization period.

CONTACTS AND LOCATIONS:
Overall Officials: Dana Portenier, MD, Principal Investigator — Duke University
Locations (1):
- Duke Regional Hospital, Durham, North Carolina, United States